CLINICAL TRIAL: NCT00323206
Title: Phase I Trial of Intratumoral pIL-12 Electroporation in Malignant Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Gene Vector Laboratory (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13224
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2009-01

CONDITIONS: Malignant Melanoma
Keywords: melanoma; electroporation; IL-12; gene therapy; gene transfer
MeSH Terms: conditions — Melanoma | interventions — Plasmids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intra-tumoral Electroporation of pIL-12 (Experimental): Participants will receive intra-tumoral injection of pIL-12 followed immediately by electrical discharge around the tumor site resulting in electroporation of plasmid DNA into tumor cells. For each lesion selected for therapy, a total of three electroporation treatments will be performed.
  Interventions: Biological: IL-12p DNA; Procedure: Intratumoral Electroporation

INTERVENTIONS:
Biological: IL-12p DNA — Plasmid IL-12 will be administered as an intratympanic (IT) injection.
  Other Names: Plasmid IL-12; pIL-12; plasmid DNA
Procedure: Intratumoral Electroporation — The electroporation apparatus with the electrical contacts will be placed around the tumor site and activated.
  Other Names: plasmid electroporation

SUMMARY:
The purpose of this research study is to study a type of gene therapy treatment called plasmid electroporation. This type of treatment involves the injection of a gene into some melanoma tumors located near the surface of the skin, followed by a burst of electricity into the tumor to cause the tumor to take up the gene. This study is a Phase I study to determine the side effects and the correct dose of this type of treatment and also its effectiveness in treating melanoma. While the electroporation technique has been used in people, the combination of plasmid injection and electroporation is being tried in human beings for the first time.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have cytologically/histologically documented metastatic malignant melanoma with lesions near the skin that would be accessible to electroporation and Fine Needle Aspiration (FNA) and biopsy.
* Age > 18 years old
* Patients must have ECOG performance status 0-2
* Patients may have had prior chemotherapy or immunotherapy (with vaccines or Interferon or IL-2) with progression or persistent disease. All chemotherapy or immunotherapy must be stopped for 4 weeks prior to electroporation. Patients may have had radiation therapy, but must have progressive disease after radiation therapy if the lesions to be electroporated are within the radiation field. In addition, it must be at least 2 weeks since administration of radiation therapy and all signs of toxicity must have abated.
* Patients must be able to give informed consent and able to follow guidelines given in the study
* Patients must have a minimum of two eligible tumors and may have up to four eligible tumors treated with electroporation.

Exclusion Criteria:

* Patients may not have had prior therapy with IL-12 or prior genetic therapy
* Patients must not have evidence of significant active infection (e.g., pneumonia, cellulitis, wound abscess, etc.) at time of study entry.
* Patients must have adequate renal and normal hepatic function (creatinine < 1.5 x upper limit of normal (ULN), bilirubin and SGOT (AST) within institutional normal limits) obtained within 4 weeks prior to registration.
* Patients must have absolute neutrophil count (ANC) > 1500/mm^3 and platelet count > 100,000 /mm^3 within 4 weeks prior to registration.
* Pregnant and breast feeding women are excluded from the study because effects on the fetus are unknown and there may be a risk of increased fetal wastage.
* Women of childbearing age must have a negative pregnancy test and be willing to use a highly effective method of contraception. Men who are sexually active must also be willing to use an accepted and effective method of contraception.
* Patients with electronic pacemakers or defibrillators are excluded from this study as the effect of electroporation on these devices is unknown. Patients with significant cardiac arrhythmia's (including ventricular tachycardia, ventricular fibrillation or WPW syndrome) are also excluded.
* Patients with a history of epilepsy are excluded unless they have been seizure free over the last 5 years and are thought to be at low risk for seizure by their neurologist.
* Tumors that invade the bone, major blood vessels or nerves are ineligible because those tumors are contraindications to the use of electroporation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 8 weeks
  MTD of intralesionally electroporated IL-12 plasmid (pIL-12) as well as a recommended dose for Phase II study. Dose-Limiting Toxicity (DLT): will be defined as hematologic toxicities or diarrhea greater than grade 3, and nonhematologic toxicities greater than grade 2 as defined in the NCI common toxicity criteria, Version 3.0. Significant local skin breakdown, cellulitis, bleeding or ulceration will preclude treatment of particular tumor nodules although treatment of other nodules can continue.

SECONDARY OUTCOMES:
Local and Systemic Response | 8 weeks
  Number of participants with tumor response.

OTHER OUTCOMES:
Local and Systemic Expression of IL-12 and IFN Gamma | 8 weeks
  Cytokine expression measured by enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Adil Daud, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: H Lee Moffiitt Cancer Center & Research Institute website — http://www.moffitt.org